CLINICAL TRIAL: NCT01900301
Title: Cholinergic Decontextualization of Exposure Therapy for Anxiety
Brief Title: Generalization of Extinction Learning
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michelle Craske, Professor, Department of Psychology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MH101359-01
Record Dates: First submitted 2013-07-08; First posted 2013-07-16 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Social Anxiety Disorder
Keywords: exposure; scopolamine; extinction learning; social anxiety
MeSH Terms: conditions — Phobia, Social | interventions — Scopolamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Scopolamine .4mg (Experimental): Participants will be randomized to either .4mg/.01 mL Scopolamine, .5mg/.01 mL Scopolamine or .6mg/.01 mL Scopolamine, administered via nasal drops, prior to each session of exposure therapy
  Interventions: Drug: Scopolamine
- Intranasal placebo (Placebo Comparator): Participants will be randomized to a placebo, administered via nasal drops, prior to each session of exposure therapy
  Interventions: Drug: intranasal placebo
- Scopolamine .5mg (Experimental): Participants will be randomized to either .4mg/.01 mL Scopolamine, .5mg/.01 mL Scopolamine or .6mg/.01 mL Scopolamine, administered via nasal drops, prior to each session of exposure therapy
  Interventions: Drug: Scopolamine
- Scopolamine .6mg (Experimental): Participants will be randomized to either .4mg/.01 mL Scopolamine, .5mg/.01 mL Scopolamine or .6mg/.01 mL Scopolamine, administered via nasal drops, prior to each session of exposure therapy
  Interventions: Drug: Scopolamine

INTERVENTIONS:
Drug: Scopolamine — Participants will be randomized to either, .4mg/.01 mL Scopolamine, .5mg/.01 mL Scopolamine or .6mg/.01 mL Scopolamine, administered via nasal drops, prior to each session of exposure therapy
  Arms: Scopolamine .4mg; Scopolamine .5mg; Scopolamine .6mg
Drug: intranasal placebo — Participants will be randomized to a drug placebo, administered via nasal drops, prior to each session of exposure therapy
  Arms: Intranasal placebo

SUMMARY:
Fear, whether it occurs in humans suffering from an anxiety disorder or in experimental models with rodents, is reduced by exposing the frightened organism to the fearful stimulus in the absence of any negative consequences (i.e., extinction, or exposure therapy). However, fear often renews when the feared stimulus is encountered in a context different from the exposure context. In rats, the investigators found that interfering with the animal's ability to process contexts during extinction by administering an anticholinergic drug prevented fear renewal. This proposal will determine if the beneficial effect of this drug translates to exposure therapy in socially anxious humans. To this end, 100 individuals with Social Phobia who fear public speaking will undergo repeated sessions of exposure to public speaking, within a virtual reality context. Participants will be randomized to either drug placebo, .4mg/.01 mL Scopolamine, .5mg/.01 mL Scopolamine or .6mg/.01 mL Scopolamine, administered via nasal drops, prior to each session of exposure therapy. One month after completion of exposure therapy, context renewal will be tested by comparing physiological and subjective responses to public speaking in the same virtual context as used during exposure therapy versus a context different than the one used during exposure therapy. The goal is to identify the dose of Scopolamine associated with the greatest reduction in context renewal. In addition, a secondary analysis will attempt to identify those individuals who benefit most from Scopolamine-augmentation of exposure therapy.

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 18 and 55,
2. fluent in English,
3. within normal body weight (BMI=18.5 to 24.9)
4. meet DSM-IV diagnostic criteria for Social Phobia and report a fear of public speaking.

Exclusion Criteria:

1. participant report of a diagnosed medical or neurological disorder
2. prescription or over the counter medications that can interact with Scopolamine, such as anticholinergic medications (e.g. belladonna alkaloids, antihistamines, meclizine, tricyclic antidepressants, and muscle relaxants), cold medicines, cough suppressants. Other drugs that will be reasons for exclusion include: antimuscarinics, nifedipine, parasympathomimetics, amantadine, amoxapine, antacids, antidiarrheals, anxiolytics, hypnotics, atomexetine, bupropion, cisapride, clozapine, cyclobenzaprine, digoxin, disopyramide, dronabinol (THC), ethanol, maprotilline, memantine, metoclopramide, nabilone, olanzapine, opiate agonists, orphenadrine, phenothiazines, potassium salts, quinidine, sedating H1-blockers, topiramate, tricyclic antidepressants, erthyromycin, ketoconazole, and tegaserod.
3. over the counter drugs or substances that may have a sedative effect (e.g. herbal sedatives: ashwagandha, Duboisia hopwoodii, Prostanthera striatiflora, kava, mandrake, valerian, cannabis, passiflora incarnate; Antihistamines: Diphenhydramine, Dimenhydrinate, Doxylamine, Promethazine; Alcohol; Dextromethorphan)
4. individuals with urinary problems (e.g., BPH)
5. pregnant or nursing females (as the effect of Scop on fetuses is not known)
6. suicidality
7. delusions or hallucinations
8. history of substance dependence in last five years or substance abuse within the past 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Eye blink startle reflex | change from final exposure session to follow-up (8 weeks following baseline)
Skin conductance responses and heart rate | change from final exposure session to follow-up (8 weeks following baseline)
Subjective Units of Distress | change from final exposure session to follow-up (8 weeks following baseline)

SECONDARY OUTCOMES:
Self Statements During Public Speaking Scale | change from baseline to follow-up (8 weeks following baseline)
Personal Report of Confidence as a Speaker Scale | change from baseline to follow-up (8 weeks following baseline)
Subjective units of distress during in vivo speech | change from baseline to follow-up (8 weeks following baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle G. Craske, Ph.D., Principal Investigator — Department of Psychology, UCLA; Michael Fanselow, Ph.D., Principal Investigator — Department of Psychology, UCLA
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Craske MG, Fanselow M, Treanor M, Bystritksy A. Cholinergic Modulation of Exposure Disrupts Hippocampal Processes and Augments Extinction: Proof-of-Concept Study With Social Anxiety Disorder. Biol Psychiatry. 2019 Nov 1;86(9):703-711. doi: 10.1016/j.biopsych.2019.04.012. Epub 2019 Apr 19. PMID 31174846